CLINICAL TRIAL: NCT04481581
Title: Titration of Inspired Oxygen During Mechanical Ventilation Using a Bedside Decision Support Tool
Brief Title: Titration of Oxygen Levels During Mechanical Ventilation With Electronic Alerts
Acronym: TOOLs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Sonal Pannu, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014H0236; 5KL2TR002734-03 (NIH)
Record Dates: First submitted 2020-06-21; First posted 2020-07-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Intervention Model Description: This will be a parallel design, unblinded, randomized (1:1) trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this study providers cannot be masked, outcome assessors and investigators will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm- Oxygen titration with electronic alerts (Experimental): Oxygen titration will be done based on electronic alerts and decisions support tool by Respiratory Therapists, if FiO2=> 0.4 and SpO2 =>94% for more than 45 minutes
  Interventions: Other: Electronic Alerts
- Control Arm- Oxygen titration by one time physician orders (No Intervention): Oxygen titration will be done ventilator management guidelines for the medical intensive care unit. Titration is done by one-time orders.

INTERVENTIONS:
Other: Electronic Alerts — When FiO2 remains =>0.4 and SpO2 =>94% for more than 45 minutes, an electronic health record based alert will be sent to respiratory therapists to titrate oxygen per decision support tool.
  Arms: Intervention arm- Oxygen titration with electronic alerts

SUMMARY:
Fractional oxygen during mechanical ventilation, is a life sustaining therapy in the intensive care unit , used for about a million patients annually. Oxygen therapy needs to be tightly balanced as both hypoxia and hyperoxia are harmful. Establishing precision in oxygenation has significant implications for improving patient outcomes, resource utilization and reducing iatrogenic harm to a vulnerable population. The investigators propose an approach using a oxygen titration protocol consisting of electronic health records based alerts to guide oxygen adjustment.

DETAILED DESCRIPTION:
The investigators will conduct a prospective randomized, clinical trial in the Medical Intensive Care Unit at Ohio State University Medical Center. In the intervention arm, respiratory therapists' will conduct oxygen titration with the help of a novel, high fidelity, electronic health records based, protocol consisting of electronic alerts and decision support tool. Oxygen titration in the control arm will be done without alerts and will be per "current standard of care".

Participants for this study will be identified and recruited from patients admitted to the Ohio State University, Wexner Medical Center and James Cancer Hospital, Medical Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

• Critically ill subjects who require mechanical ventilation for at least 24 hours.

Exclusion Criteria:

* Subjects without research authorization,
* Pregnancy,
* Pneumothorax,
* Carbon monoxide poisoning,
* Hyperbaric oxygen therapy
* Acute ST elevation Myocardial Infarction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Duration of Hyperoxemia | Duration of Mechanical Ventilation, an average of 10-14 days
  The degree of excess exposure will be recorded as percent FiO2 >0.4 when saturation continued to remain above 94%. Primary outcome will be determined by the proportion of time the patient will be "exposed to excessive supplied oxygen" divided by the total time under mechanical ventilation.

SECONDARY OUTCOMES:
Ventilator Free days | 28 days
  The number of days between successful weaning from mechanical ventilation and day 28 after study enrollment.
ICU length of stay | days of ICU stay within hospitalization, average of 20-25 days
  Duration of stay in the intensive care unit after patient enrollment
Duration of stay in the hospital after patient enrollment | Current Hospital Stay, upto 30 days
  Duration of stay in the hospital after patient enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sonal R Pannu, M.D., Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pannu SR, Haddad T, Exline M, Christman JW, Horowitz JC, Peters J, Brock G, Diaz P, Crouser ED. Rationale and design of a randomized controlled clinical trial; Titration of Oxygen Levels (TOOL) during mechanical ventilation. Contemp Clin Trials. 2022 Aug;119:106811. doi: 10.1016/j.cct.2022.106811. Epub 2022 May 31. PMID 35660485